CLINICAL TRIAL: NCT06361420
Title: The Efficacy of Driving Pressure-guided Lung Protective Ventilation in Surgical Repair of Acute Type A Aortic Dissection: an Open-label, Randomized Control Clinical Trial
Brief Title: Driving Pressure-guided Lung Protective Ventilation
Acronym: DPV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Lin, PhD (Other)
Responsible Party: Sponsor-Investigator, Yong Lin, PhD, Associate chief physician, Fujian Medical University Union Hospital
Organization: Fujian Medical University Union Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023YF051-01
Record Dates: First submitted 2024-03-10; First posted 2024-04-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypoxemia; Ventilator Lung
Keywords: Driving Pressure; Lung Protective Ventilation; Aortic Dissection; Hypoxia; Postoperative Pulmonary Complications
MeSH Terms: conditions — Hypoxia; Aortic Dissection

STUDY DESIGN:
Intervention Model Description: open, randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Driving pressure-guided lung protective ventilation during the surgery (Experimental): A 10-cycle experimental ventilation will be carried out at each level of positive end expiratory pressure after intubation, and the driving pressure of the last cycle will be recorded. The positive end expiratory pressure value corresponding to the lowest driving pressure is recognised as the optimal ventilation parameter.
  Interventions: Procedure: Driving pressure-guided positive end expiratory pressure; Procedure: Ventilation strategy; Procedure: Management of hypoxemia
- Conventional lung protective ventilation (Other): Positive end expiratory pressure will be maintained at the level facilitating optimal oxygenation during the off-pump period.
  Interventions: Procedure: Optimal oxygenation-guided positive end expiratory pressure; Procedure: Ventilation strategy; Procedure: Management of hypoxemia

INTERVENTIONS:
Procedure: Driving pressure-guided positive end expiratory pressure — The positive end expiratory pressure setting rules are as follows: a 10-cycle experimental ventilation will be carried out at each level of positive end expiratory pressure after intubation, and the driving pressure of the last cycle will be recorded. The positive end expiratory pressure value corresponding to the lowest driving pressure is recognised as the optimal ventilation parameter. Partial pressure of carbon dioxide monitoring is employed to determine the tidal volume and respiratory rate. Inspiration/expiration pattern is adjusted based on the preoperative small airway condition. This parameter is subject to modification upon cessation of ventilation, ICU admission, and every morning throughout the ventilation period. During cardiopulmonary bypass, mechanical ventilation is maintained using the low-level parameters.
  Arms: Driving pressure-guided lung protective ventilation during the surgery
Procedure: Optimal oxygenation-guided positive end expiratory pressure — Positive end expiratory pressure will be maintained at the level facilitating optimal oxygenation during the off-pump period. Partial pressure of carbon dioxide monitoring is employed to determine the tidal volume and respiratory rate. Inspiration/expiration pattern is adjusted based on the preoperative small airway condition. This parameter is subject to modification upon cessation of ventilation, ICU admission, and every morning throughout the ventilation period. During cardiopulmonary bypass, mechanical ventilation is maintained using the low-level parameters.
  Arms: Conventional lung protective ventilation
Procedure: Ventilation strategy — A Pressure regulated volume control mode is used in the patients before extubation. The ventilation target are: (1) a pulse oximetry ≥ 90% or a partial pressure of arterial oxygen ≥ 60mm Hg; (2) a partial pressure of arterial carbon dioxide: 35 ~ 50 mm Hg and (3) a pondus hydrogenii (pH) value > 7.20. The ventilation parameters are: (1) tidal volume: 6 ~ 8 mL/Kg predictive body weight; (2) respiratory rate 10 ~ 15 cycles per minute; (3) inspiratory/expiratory ratio: 1:1.5 (1:2.5 - 1:3 in the patients with chronic obstructive pulmonary disease); positive end expiratory pressure: 0 ~ 8 cm centimeter water column. On-pump ventilation parameters are: (1) tidal volume: 4 mL/Kg predictive body weight; (2) respiratory rate: 4 circles per minute; (3) positive end-expiratory pressure: 4 cm centimeter water column; (4) inspiratory oxygen fraction: 21%.
  Other Names: Same part of ventilation strategy between the two groups
Procedure: Management of hypoxemia — Management of hypoxemia will be initiated immediately through the following steps: (1) carefully checking anaesthesia apparatus malfunction, airway normality, and monitoring accuracy; (2) improving cardiac function, correcting fluid overload, and alleviating systemic inflammation; (3) performing alveolar recruitment manoeuvres as described above; (4) increasing the tidal volume and positive end expiratory pressure within the upper limits; (5) increasing the respiratory rate while addressing concurrent hypercapnia; (6) titrating the fraction of inspiratory oxygen until the pulse oximetry reaches or exceeds 90%; and (7) considering the use of extracorporeal membrane oxygenation if any following situations occurred 14: (a) a partial pressure of arterial oxygen < 50 mm Hg for more than 3 hours; (b) a partial pressure of arterial oxygen to inspiratory oxygen fraction ratio < 80 mm Hg for more than 6 hours; or (c) a critical respiratory acidosis for more than 6 hours.

SUMMARY:
The study, named as "The Efficacy of Driving Pressure-guided Lung Protective Ventilation in Surgical Repair of Acute Type A Aortic Dissection: an open-label, randomized control clinical trial", aims to investigate whether driving pressure-guided lung protective ventilation can reduce postoperative oxygenation function in patients who have undergone surgical repair of acute type A aortic dissection. The primary outcomes is the incidence of postoperative hypoxemia (a partial pressure of arterial oxygen to inspiratory oxygen fraction ratio less than 300 mm Hg or a peripheral blood oxygen saturation less than 93% at any concentration of inspiratory oxygen) within 7 days after the surgery.

DETAILED DESCRIPTION:
Postoperative hypoxemia is defined as a partial pressure of arterial oxygen to inspiratory oxygen fraction ratio less than 300 mm Hg or a peripheral blood oxygen saturation less than 93% at any concentration of inspiratory oxygen. Acute type A aortic dissection is a lethal disease requiring emergency surgery. Compared with non-cardiac surgery, hypoxemia frequently occurs after surgical repair for acute type A aortic dissection which has been reported to be 52%-67.6%, and the possible mechanisms are as followed: (1) systemic inflammatory reaction induced by massive thrombosis formation and long duration of extracorporeal circulation; (2) ischemia-perfusion injury in lung; and (3) a massive perioperative transfusion. Postoperative hypoxemia has been reported to be associated with prolonged duration of extubation, length of stay in ICU and respiratory failure, which contributes a high mortality of 20% to 44%.

Driving pressure, defined as the difference between platform airway pressure and positive end-expiratory pressure, was first introduced by Amato and his colleagues in their meta-analysis study on acute respiratory distress syndrome in 2015, demonstrating that driving pressure was most strongly associated with survival among various ventilation parameters. A lower driving pressure has been verified to be closely relative to an ameliorative prognosis after surgery. However, controversy persists regarding whether driving pressure-guided ventilation can decrease the incidences of postoperative hypoxemia and other pulmonary complications in the patients underwent surgical repair of acute type A aortic dissection.

Given the need for additional evidence to confirm the relationship between driving pressure and postoperative hypoxemia in the patients with acute type A aortic dissection, this open-label, randomized control clinical trial aims to assess the efficacy and safety of the driving pressure-guided lung protective ventilation strategy in preventing hypoxemia and other pulmonary complications after the surgical repair for acute type A aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Able to sign Informed Consent and Release of Medical Information Forms;
2. Age ≥ 14 years and ≤ 70 years old;
3. Being confirmed the diagnosis by chest computed tomography angiography and receiving the surgical repair of acute type A aortic dissection.

Exclusion Criteria:

1. Age < 14 years or > 70 years old;
2. Sepsis before surgery;
3. Chronic pulmonary disease including lung infection or asthma requiring long-term pharmacotherapy;
4. History of lung tumor;
5. Obstructive sleep apnea hypopnea syndrome requiring long-term noninvasive mechanical ventilation support;
6. Heart failure requiring catecholamines or invasive mechanical ventilation support;
7. Body mass index > 30 Kg·m-2;
8. Being reluctance to participate this study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative hypoxemia | Within 7 days after surgery
  Postoperative hypoxemia is defined as a partial pressure of arterial oxygen to inspiratory oxygen fraction ratio less than 300 mm Hg or a pulse oximetry less than 93% at any concentration of inspiratory oxygen that occurred from admission to the operating room to 7 days post-surgery.

SECONDARY OUTCOMES:
The trend of perioperative oxygenation function | Within 7 days after surgery
  An automated blood gas analyzer will be applied for arterial blood gas analyses, with the time points: T1 (before surgery), T2 (after intubation), T3 (withdrawal from cardiopulmonary bypass), T4 (end of surgery), T5 (postoperative day 1), T6 (postoperative day 3), T7 (postoperative day 5), and T8 (postoperative day 7).
Postoperative pulmonary complications except hypoxemia | Within 7 days after surgery
  Postoperative pulmonary complications are defined as any postoperative respiratory system complication that occurs from admission to the intensive care unit to 7 days post-surgery, encompassing (1) respiratory infection, (2) respiratory failure, (3) bronchospasm, (4) atelectasis, (5) pleural effusion, (6) pneumothorax, and (7) aspiration pneumonitis.
Early/late death | Within 30 days after surgery
  Early death was defined as any death occurring within 72 hours of surgery, while late death was considered for deaths occurring within 30 days after the surgery was scheduled.
Vasoactive-inotropic score at the end of surgery | Within 7 days after surgery
  The vasoactive-inotropic score is the sum of the dosages of frequently used vasoactive or inotropic agents according to the weighted values of the enrolled patients. Vasoactive-Inotropic Score = dopamine dose (μg·kg-1·min-1) + dobutamine dose (μg·kg-1·min-1) + 100 × epinephrine dose (μg·kg-1·min-1) + 10 × phosphodiesterase inhibitor (milrinone or olprinone) dose (μg·kg-1·min-1) + 100 × norepinephrine dose (μg·kg-1·min-1) +10000 × vasopressin dose (U·kg-1·min-1).
Postoperative adverse cardiovascular events | Within 7 days after surgery
  The postoperative adverse cardiovascular events include new-onset lethal arrhythmias (supraventricular/ventricular tachycardia, ventricular fibrillation, or Adams-Stokes syndrome), acute myocardial infarction, cardiogenic shock, and thrombotic or embolic events.
Length of stay in intensive care unit | Within 30 days after surgery
  The duration from admission to discharge of the ICU
Ventilation assistance time | Depending on the time point of extubation, not exceeding 30 days
  Duration from the end of the surgery to extubation.
Postoperative extrapulmonary complications | Within 7 days after surgery
  Postoperative extrapulmonary complications include tracheotomy, rethoracotomy for exploration, wound infection, sepsis, gastrointestinal haemorrhage, and neurological complications (such as delayed recovery, delirium, cognitive dysfunction, coma, new-onset stroke, and syncope)

CONTACTS AND LOCATIONS:
Overall Officials: Yong Lin, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian medical university union hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No